CLINICAL TRIAL: NCT02411929
Title: A Phase 1, Open-Label, Non-Randomized, 2-Period, Fixed Sequence, Study to Assess the Absolute Bioavailability and Fraction Absorbed of Ertugliflozin in Health Male Subjects Using a 14^C-Microdose Approach
Brief Title: A Phase 1 Study of Ertugliflozin in Healthy Male Participants (MK-8835-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8835-020; B1521043 (Other: Pfizer Protocol Number)
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ertugliflozin (Experimental): Period 1: Oral dose of 15 mg unlabeled ertugliflozin + intravenous (IV) dose of 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C. The 14^C IV dose will be administered as an infusion over approximately 5 minutes starting at 55 minutes after the unlabeled oral dose. → Period 2: Oral dose 15 mg unlabeled ertugliflozin + oral dose of 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C. Both the unlabeled and 14^C-ertugliflozin will be administered at the same time (no more than 5 minutes apart). Dosing in Periods 1 and 2 will be separated by a washout of at least 11 days.
  Interventions: Drug: Unlabeled ertugliflozin for oral use; Drug: 14^C-labeled ertugliflozin for IV use; Drug: 14^C-labeled ertugliflozin for oral use

INTERVENTIONS:
Drug: Unlabeled ertugliflozin for oral use — 15 mg oral (3 x 5 mg tablets)
Drug: 14^C-labeled ertugliflozin for IV use — 100 µg (10 µg/mL solution IV) containing approximately 400 nCi 14^C (ie, radiolabeled ertugliflozin)
Drug: 14^C-labeled ertugliflozin for oral use — 100 µg (10 µg/mL solution oral) containing approximately 400 nCi 14^C (ie, radiolabeled ertugliflozin)

SUMMARY:
This study will evaluate the absolute oral bioavailability (F) and fraction absorbed (Fa) of ertugliflozin following oral administration of unlabeled ertugliflozin (MK-8835) and intravenous (IV) and oral administration of 14^C-labeled ertugliflozin in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 65 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs.)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies).
* Any clinically significant malabsorption condition (eg, gastrectomy, bowel resection).
* A positive urine drug screen for drugs of abuse or recreational drugs.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
* History of abuse of alcohol or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Current smokers and those who have smoked any substance within the last 12 months.
* Treatment with an investigational drug within 1 month preceding the first dose of study medication.
* Have participated in any clinical study with exposure to 14^C in the last 12 months.
* Any radiation exposure, including that which is projected to result from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures. No occupationally exposed worker, as defined in the Ionising Radiation Regulation 1999, shall participate in the study.
* Use of prescription or nonprescription drugs (including vitamins and dietary supplements) within 7 days prior to the first dose of study medication.
* Use of herbal supplements within 28 days prior to the first dose of study medication.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* Participants who have previously participated in a clinical trial for ertugliflozin.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Raje S, Callegari E, Sahasrabudhe V, Vaz A, Shi H, Fluhler E, Woolf EJ, Schildknegt K, Matschke K, Alvey C, Zhou S, Papadopoulos D, Fountaine R, Saur D, Terra SG, Stevens L, Gaunt D, Cutler DL. Novel Application of the Two-Period Microtracer Approach to Determine Absolute Oral Bioavailability and Fraction Absorbed of Ertugliflozin. Clin Transl Sci. 2018 Jul;11(4):405-411. doi: 10.1111/cts.12549. Epub 2018 Mar 25. PMID 29575530
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Ertugliflozin
Started | 8
Completed | 8
Not Completed | 0
Period: Washout Period
Arm/Group | Ertugliflozin
Started | 8
Completed | 8
Not Completed | 0
Period: Period 2
Arm/Group | Ertugliflozin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ertugliflozin
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUC Last) (Dose Normalized to 1 mg) and Absolute Oral Bioavailability (F) (Period 1)
Description: AUC0-inf is a measure of the mean concentration levels of drug in the plasma after the drug dose. An absolute bioavailability provides information on the amount of a drug reaching the systemic circulation and can be determined by comparing the plasma concentration-time-curves (area under the curve) of a compound after oral application of that compound to that after intravenous application of the same compound.
Time Frame: Oral: 0, 15 and 30 min., and at 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs. after oral dose; IV: -5 min. (predose), 0 (end of infusion), and at 10, 20, 30, and 45 min. and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 11, 23, 47, 71, and 95 hrs. after end of infusion
Population: The pharmacokinetic (PK) Parameter Analysis Population for ertugliflozin is defined as all participants treated who have at least 1 of the ertugliflozin PK parameters of interest. The PK Parameter Analysis Population for 14^C-ertugliflozin analysis is defined as all participants treated who have at least 1 of the 14^C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: AUCinf(dn), ng•hr/mL/mg
Groups:
- Unlabeled Ertugliflozin 15 mg Oral: Oral dose of 15 mg unlabeled ertugliflozin on Day 1 of Period 1
- 14^C-Ertugliflozin 100 ug IV: 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C IV administered as an infusion over approximately 5 minutes starting at 55 minutes after the unlabeled oral dose on Day 1 of Period 1.
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 8
AUCinf(dn), ng•hr/mL/mg | 93.16 (13) | 88.96 (15)
Statistical Analysis 1: Comparison: Unlabeled Ertugliflozin 15 mg Oral vs 14^C-Ertugliflozin 100 ug IV; Ratio - Test (oral) / Reference (IV) of means; Test type: Superiority or Other; Test (oral)/Reference (IV) of means = 104.73, 90% CI 2-sided [101.64 to 107.91] — Natural log transformed AUCinf(dn) and AUClast(dn) from Period 1 were analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences were exponentiated

2. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUC Last) Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug IV (Period 1) (Dose Not Normalized to 1 mg)
Description: AUC0-last is a measure of the total amount of drug in the plasma from time zero to time of the last measurable concentration. Geometric coefficient of variation is given as the percent coefficient of variation.
Time Frame: as for outcome 1
Population: The PK Parameter Analysis Population for ertugliflozin is defined as all participants treated who have at least 1 of the ertugliflozin PK parameters of interest. The PK Parameter Analysis Population for 14^C-ertugliflozin analysis is defined as all participants treated who have at least 1 of the 14^C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 8
ng•hr/mL | 1376 (12) | 7.859 (14)

3. Secondary Outcome: Pharmacokinetic Parameter: (AUC Inf) Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: AUC0-inf is a measure of the mean concentration levels of drug in the plasma after the dose. Geometric coefficient of variation is given as the percent coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 8
ng•hr/mL | 1397 (13) | 8.477 (15)

4. Secondary Outcome: Pharmacokinetic Parameter: Maximum Plasma Concentration (Cmax) Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1) (Dose Normalized to 1 mg)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Geometric coefficient of variation is given as the percent coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 8
ng/mL/mg | 17.09 (14) | 89.34 (32)

5. Secondary Outcome: Pharmacokinetic Parameter: Time for Cmax (Tmax) Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. The confidence intervals displayed are minimums to maximums.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 8
Hours | 1.00 [1.00 to 1.50] | 0.083 [0.083 to 0.100]

6. Secondary Outcome: Pharmacokinetic Parameter: Terminal Elimination Half-Life (t1/2) Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 8
Hours | 14.04 (2.17) | 8.098 (2.248)

7. Secondary Outcome: Pharmacokinetic Parameter: Apparent Oral Total Plasma Clearance (CL/F) - Oral, Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: Apparent clearance is a calculation of the rate at which a drug is removed from plasma after oral administration via renal, hepatic and other clearance pathways, expressed as volume (milliliters) per unit of time (minutes). Geometric coefficient of variation is given as the percent coefficient of variation. This outcome measure is for the Ertugliflozin oral drug profile only so no participants were analyzed in the 14^C-Ertugliflozin 100 ug IV arm.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min.
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 0
mL/min. | 178.7 (13) |

8. Secondary Outcome: Pharmacokinetic Parameter: Systemic IV Total Plasma Clearance (CL) - IV, Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: Systemic clearance is a calculation of the rate at which a drug is removed from plasma via renal, hepatic and other clearance pathways, expressed as volume (milliliters) per unit of time (minutes). Geometric coefficient of variation is given as the percent coefficient of variation. This outcome measure is for the Ertugliflozin intravenous drug profile only so no participants were analyzed in the Ertugliflozin oral arm.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min.
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 0 | 8
mL/min. |  | 187.2 (15)

9. Secondary Outcome: Pharmacokinetic Parameter: Apparent Volume of Distribution (Vz/F) Following Oral Administration - Oral, Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose is influenced by the fraction absorbed. Geometric coefficient of variation is given as the percent coefficient of variation. This outcome measure is for the Ertugliflozin oral drug profile only so no participants were analyzed in the 14^C-Ertugliflozin 100 ug intravneous arm.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 8 | 0
Liters | 215.3 (21) |

10. Secondary Outcome: Pharmacokinetic Parameter: Steady-State Volume of Distribution (Vss) Following IV Infusion - IV, Following Administration of Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ertugliflozin 100 ug IV (Period 1)
Description: Steady-State Volume of Distribution is the theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it is in blood plasma at steady state. Geometric coefficient of variation is given as the percent coefficient of variation. This outcome measure is for the Ertugliflozin intravenous drug profile only so no participants were analyzed in the Ertugliflozin oral arm.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 0 | 8
Liters |  | 85.53 (15)

11. Secondary Outcome: Pharmacokinetic Parameter: Fraction Absorbed (Fa, Radioactivity in Urine) (Periods 1 and 2) (Dose Normalized)
Description: Fraction absorbed is the fraction of the total ertugliflozin dose absorbed, regardless of the fate of that dose after absorption (i.e., metabolism, degradation, etc). Fraction Absorbed was estimated as the ratio of total radioactivity (dose normalized) excreted into the urine (from time zero to the time of last measurable concentration) following oral and IV administration of 14^C-ertugliflozin. Fraction of 14^C dose recovered in urine = 14^C total in urine in dpm/14^C total in dose in dpm
Time Frame: Part 1: pre- IV dose, 0-11 and 11-23 hrs. post IV dose, and 23 - 47, 47 - 71 and 71 - 95 hrs. until Day 5; Part 2: predose, 0-12 and 12-24 hrs. post dose, and then 24-hour intervals until Day 5
Population: The estimated Fa Population included only the 6 participants with complete urine data for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction of 14^C dose recovered in urine
Groups:
- 14^C-Ertugliflozin 100 ug Oral: 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C administered orally after the unlabeled oral dose (no more than 5 minutes apart) on Day 1 of Period 2.
Arm/Group | 14^C-Ertugliflozin 100 ug Oral | 14^C-Ertugliflozin 100 ug IV
Number analyzed (Participants) | 6 | 6
Fraction of 14^C dose recovered in urine | 0.432 (10) | 0.390 (19)
Statistical Analysis 1: Comparison: 14^C-Ertugliflozin 100 ug Oral vs 14^C-Ertugliflozin 100 ug IV; Ratio - Test (Oral) / Reference (IV) (%); Test type: Superiority or Other; Ratio = 110.71 — The ratio (Test/Reference) of the geometric means of dose normalized natural log transformed Total 14^C in Urine will be estimated. Total 14^C_Urine_IV is the Reference formulation and Total 14C_Urine_Oral is the Test formulation (expressed as a %)

12. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (Periods 1 and 2)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 33 days
Population: The Safety Population included all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug IV: Period 1: Oral dose of 15 mg unlabeled ertugliflozin + intravenous (IV) dose of 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C. The 14^C IV dose will be administered as an infusion over approximately 5 minutes starting at 55 minutes after the unlabeled oral dose.
- Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug Oral: Period 2: Oral dose 15 mg unlabeled ertugliflozin + oral dose of 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C. Both the unlabeled and 14^C-ertugliflozin will be administered at the same time (no more than 5 minutes apart).
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug IV | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug Oral
Number analyzed (Participants) | 8 | 8
Participants | 3 | 1

13. Secondary Outcome: Number of Participants Discontinuing Study Drug Due to Adverse Events (Periods 1 and 2)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 16 days
Population: The Safety Population included all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug IV | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug Oral
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 33 days
Description: The Safety Population included all participants who received at least one dose of study drug.
Groups:
- Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug Oral: Period 2: Oral dose 15 mg unlabeled ertugliflozin + oral dose of 100 µg 14^C-labeled ertugliflozin containing approximately 400 nCi 14^C. Both the unlabeled and 14^C-ertugliflozin will be administered at the same time (no more than 5 minutes apart.)
Arm/Group | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug IV | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug Oral
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug IV (N=8) | Unlabeled Ertugliflozin 15 mg Oral + 14^C-Ert. 100 ug Oral (N=8)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation) to the sponsor at least 30 days before they are submitted for publication or otherwise disclosed. An additional 60 days will be requested if any patent action is required to protect intellectual property rights. The investigator will, on request, remove any previously undisclosed confidential information before disclosure.